CLINICAL TRIAL: NCT06266104
Title: Image Enhanced Endoscopy Technology to Improve the Detection of Colorectal Dysplasia in Patients With Inflammatory Bowel Disease
Brief Title: Image Enhanced Endoscopy IBD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Royal Perth Hospital (Other)
Responsible Party: Principal Investigator, Sherman Picardo, Doctor, Principal Investigator, Royal Perth Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: Protocol V1.4_04012024
Record Dates: First submitted 2024-02-04; First posted 2024-02-20 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Inflammatory Bowel Diseases; Dysplasia
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dye Spray Chromoendoscopy (Placebo Comparator): Patients undergoing surveillance with dye spray chromoendoscopy
  Interventions: Procedure: Image Enhanced Endoscopy Filters
- TXI (Active Comparator): Patients undergoing surveillance with TXI (Texture and Colour Enhancement Imaging)
  Interventions: Procedure: Image Enhanced Endoscopy Filters
- LCI (Active Comparator): Patients undergoing surveillance with LCI (Linked Colour Imaging )
  Interventions: Procedure: Image Enhanced Endoscopy Filters

INTERVENTIONS:
Procedure: Image Enhanced Endoscopy Filters — Patients that undergoing surveillance and consent to be involved in the study will be randomised to undergo surveillance with LCI, TXI or dye-spray chromoendoscopy (methylene blue).

SUMMARY:
Dye- spray chromoendoscopy remains the recommended gold standard approach for IBD dysplasia surveillance colonoscopy however recently published European and American guidelines recommend either dye-spray or virtual chromoendoscopy can be used for surveillance. The newer Imaged Enhanced Endoscopy technologies TXI and LCI have not formally been evaluated in IBD surveillance in a randomised controlled trial setting. These modes can easily be applied during colonoscopy and if demonstrated to be effective may save time and eliminate the need for dye-spray chromoendoscopy in the future.

ELIGIBILITY:
Inclusion Criteria:

* Patients with inflammatory bowel disease aged 18 to 75 years, that meet Australian recommendations to undergo surveillance colonoscopy will be identified and invited participate in the study.

Exclusion Criteria:

* Any active disease
* Inadequate bowel preparation
* Previous surgical resection involving the colon
* History of bowel cancer

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2024-04-03 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Dysplasia Detection Rate | 2 years
  Overall Dysplasia Detection rate

SECONDARY OUTCOMES:
Withdrawal times | 2 years
  Withdrawal time for procedure
Characterisation of lesions | 2 years
  Accurate characterisation compared to histology

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Perth Hosptial, Perth, Western Australia, Australia

IPD SHARING:
Plan to Share IPD: No